CLINICAL TRIAL: NCT06661941
Title: Predictive Tools for the Presence of Significant Coronary Artery Disease Requiring Intervention in Chronic Hemodialysis Patients
Acronym: CAD in HD
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Thana Thongsricome, MD, Thana Thongsricome, MD, Chulalongkorn University
Other Study IDs: 0042/65
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Hemodialysis; Coronary Arterial Disease (CAD); ESRD (End Stage Renal Disease)
Keywords: hemodialysis; coronary artery disease; electrocardiography; echocardiography; troponin; coronary angiography
MeSH Terms: conditions — Renal Insufficiency, Chronic; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Positive coronary artery disease: Presence of significant coronary artery disease requiring intervention from a coronary angiography result
- Negative coronary artery disease: Absence of significant coronary artery disease requiring intervention from a coronary angiography result

SUMMARY:
Medical record data of all HD patients undergoing coronary angiography (CAG) at King Chulalongkorn Memorial Hospital between January 2017 and March 2021 were retrospectively reviewed as a discovery cohort to identify factors discriminating patients with and without significant CAG-established CAD. HD patients receiving CAG between April 2021 and March 2023 were assigned as a validation cohort.

DETAILED DESCRIPTION:
Background: Hemodialysis (HD) patients have increased cardiovascular risk. Coronary artery disease (CAD) may not typically manifest in these patients and the investigational results can be confounded by the fluctuation of body fluid and electrolytes. This study explored the accuracy of these findings in identifying CAD in HD patients.

Methods: Medical record data of all HD patients undergoing coronary angiography (CAG) at King Chulalongkorn Memorial Hospital between January 2017 and March 2021 were retrospectively reviewed as a discovery cohort to identify factors discriminating patients with and without significant CAG-established CAD. HD patients receiving CAG between April 2021 and March 2023 were assigned as a validation cohort.

ELIGIBILITY:
Inclusion Criteria:

* All adult HD patients undergoing CAG at King Chulalongkorn Memorial Hospital of all indications between January 2017 and March 2021 with complete data

Exclusion Criteria:

* Those resinged for using their clinical data for the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult HD patients undergoing CAG at King Chulalongkorn Memorial Hospital of all indications between January 2017 and March 2021 with complete data
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Presence of coronary artery disease | Any positive result between January 2017 and March 2023
  Presence of significant coronary artery disease requiring intervention from a coronary angiography result

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Patient confidential data

REFERENCES:
- [Background] Go AS, Bansal N, Chandra M, Lathon PV, Fortmann SP, Iribarren C, Hsu CY, Hlatky MA; ADVANCE Study Investigators. Chronic kidney disease and risk for presenting with acute myocardial infarction versus stable exertional angina in adults with coronary heart disease. J Am Coll Cardiol. 2011 Oct 4;58(15):1600-7. doi: 10.1016/j.jacc.2011.07.010. PMID 21958887